CLINICAL TRIAL: NCT05888246
Title: Measuring the Range of Cardiac Magnetic Parameters in Healthy Subjects by Magnetocardiogram: a Prospective, Observational Clinical Study
Brief Title: Measuring the Range of Cardiac Magnetic Parameters in Healthy Subjects by Magnetocardiogram
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Nuochi Life Science Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Hangzhounuochi
Record Dates: First submitted 2022-06-29; First posted 2023-06-05 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Healthy People

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic test (Experimental): Diagnostic test: magnetocardiogram.
  Interventions: Diagnostic Test: Magnetocardiogram

INTERVENTIONS:
Diagnostic Test: Magnetocardiogram — Magnetocardiogram consists of acquisition and control system (including software) and detection part. Acquisition and control system mainly includes: cabinet, display, host, sensor. The detection part mainly includes: inspection bed, array sensor support frame, magnetic shielding equipment.

SUMMARY:
A prospective and observational clinical study of measuring the range of cardiac magnetic parameters in healthy people with the magnetocardiogram manufactured by Hangzhou Nuochi Life Science Co., LTD

DETAILED DESCRIPTION:
This study is a prospective and observational study on the collection of cardiac magnetic signals from healthy subjects by magnetocardiogram. It is expected that 412 subjects will be examined by magnetocardiography, and the range of parameters related to magnetocardiography in healthy subjects will be reported.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy people aged 18-70 years old;
2. Subjects receiving physical examination in physical examination institutions, or in other departments other than heart disease (such as orthopedics, gynecology, etc.), or in cardiology department, excluded from coronary heart disease;
3. No history of coronary heart disease;
4. ECG did not indicate myocardial ischemia or infarction;
5. Sinus rhythm without arrhythmia;
6. The subject or the subject's legal representative has been informed of the nature of the study, understands the purpose of the clinical study, voluntarily participates in the study and signs the informed consent.

Exclusion Criteria:

1. Acute coronary syndrome requires emergency PCI treatment, and it is estimated that magnetic cardiogram examination will affect the timing of emergency PCI surgery;
2. Subjects with metal implants in the thoracic cavity (including the heart cavity), such as those who have received pacemaker therapy or cardiac resynchronization therapy (CRT, CRT-D) or implantable cardioverter defibrillator (ICD) implantation, or those who have received metal heart valve implantation;
3. There is hemodynamic instability, which is defined as systolic blood pressure < 80mmHg, or cardiogenic shock; Or need vasoactive drug therapy; Intra-aortic balloon counterpulsation may be required; Or other hemodynamic support devices; As syndrome;
4. Severe tachycardia (ventricular rate > 150 beats/min), ventricular flutter, ventricular fibrillation and other malignant arrhythmias;
5. Subjects unable to lie flat (supine position);
6. Subjects with mental illness, unconscious or uncontrollable ability; Or claustrophobic subjects;
7. Other circumstances in which the investigator considers the subject inappropriate for participation in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2022-05-07 (Actual); Primary Completion 2022-05-14 (Actual); Study Completion 2022-05-14 (Actual)

PRIMARY OUTCOMES:
PR interval | 24 hours
  PR interval is defined as the position from the starting point of P wave to the starting point of QRS wave after the superposition of 36 channels in the magnetocardiogram (butterfly diagram).
QRS interval | 24 hours
  QRS interval is defined as the time (ms) from the beginning of QRS to the end of QRS after the stacking of 36 channels in the magnetocardiogram (butterfly diagram).
QT interval | 24 hours
  QT interval is defined as the time (ms) from the beginning of Q wave to the end of T wave after the stacking of 36 channels in the magnetocardiogram (butterfly diagram).
Corrected QT interval | 24 hours
  The corrected QT interval was defined as the QTC interval (ms) after the stacking of 36 channels in the magnetocardiogram (butterfly diagram). QTc = QT/(RR^0.5), RR is the average RR interval calculated by cardiac magnetic waveform, QT is QT interval.
The magnetic field intensity parameter (R/T ratio) | 24 hours
  The magnetic field intensity parameter (R/T ratio) is defined as the ratio of the maximum magnetic field intensity of the r-wave vertex to the T-wave vertex of the magnetocardiogram calculated based on the isomagnetic map.
Maximum current vector angle (MCV angle) | 24 hours
  The Angle of the maximum current vector was measured at the vertex of QRS and T wave respectively.
Maximum current vector amplitude (MCV amplitude) | 24 hours
  The amplitude of the maximum current vector was measured at the vertex of QRS wave and T wave respectively.
Total current vector angle (TCV angle) | 24 hours
  TCV represents the total current vector, which is the sum of all current vectors of 36 channels in the magnetocardiogram. First calculate the vector sum of the 36 channels, and finally calculate the angles.
Total current vector amplitude (TCV amplitude) | 24 hours
  TCV represents the total current vector, which is the sum of all current vectors of 36 channels in the magnetocardiogram. First calculate the vector sum of the 36 channels, and finally calculate the amplitude.

CONTACTS AND LOCATIONS:
Overall Officials: Jianan Wang, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No